CLINICAL TRIAL: NCT02128191
Title: Efficacy and Safety of No Treatment Compared With Oral Ibuprofen Treatment for Patent Ductus Arteriosus in Preterm Infants: a Randomized, Double-blind, Placebo-controlled, Non-inferiority Clinical Trial
Brief Title: No Treatment Versus Oral Ibuprofen Treatment for Patent Ductus Arteriosus in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se In Sung, M.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-07-129
Record Dates: First submitted 2014-04-23; First posted 2014-05-01 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Bronchopulmonary Dysplasia (BPD)
Keywords: Patent ductus arteriosus; Ibuprofen; Bronchopulmonary dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Ductus Arteriosus, Patent | interventions — Ibuprofen; Long-Term Synaptic Depression; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral ibuprofen (Active Comparator): Initial dose of 10 mg/kg of oral ibuprofen, followed by 2 doses of 5 mg/kg 24 and 48 h later
  Interventions: Drug: Oral ibuprofen
- Normal saline (Placebo Comparator): Initial dose of normal saline followed by second and third dose 24 and 48 hours later, at equal volume to ibuprofen arm
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Oral ibuprofen — Initial dose of 10 mg/kg of oral ibuprofen, followed by two doses of 5 mg/kg 24 and 48 hours later
  Other Names: Brufen® syrup, Samil pharm. Co., Ltd.
  Arms: Oral ibuprofen
Drug: Normal saline — Initial dose of normal saline followed by second and third dose 24 and 48 hours later, at equal volume to ibuprofen arm
  Other Names: Sodium chloride, Huons. Inc.
  Arms: Normal saline

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of no treatment compared with ibuprofen treatment for patent ductus arteriosus in preterm infants. The study hypothesis is that no treatment is not inferior to oral ibuprofen treatment in preterm infants. (non-inferiority study)

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, non-inferiority clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age of 30 weeks or less or birth weight of 1250 g or less
2. born in Samsung Medical Center
3. confirmed to have hemodynamically significant patent ductus arteriosus (PDA) during day of life (DOL) 5 to 14
4. Definition of hemodynamically significant PDA: ductal size ≥ 1.5 mm with left-to-right shunt (or bidirectional shunt with dominant left-to-right blood flow) on the initial echocardiography plus at least one of clinical criteria.

   * Clinical criteria

     * Respiratory signs, including tachypnea, chest retraction, increased respiratory support, unable to wean respiratory support
     * Physical signs, including a murmur, hyperdynamic precordium or bounding pulses
     * Blood pressure problems, including decreased mean or diastolic pressure or increased pulse pressure
     * Signs of congestive heart failure, including cardiomegaly, hepatomegaly or pulmonary congestion

Exclusion Criteria:

* Mortality within the first 48 hours of life
* Ductal size < 1.5 mm on the initial echocardiography
* Right-to-left shunt or bidirectional shunting with dominant right-to-left shunt through PDA
* congenital anomaly
* bilateral intraventricular hemorrhage of grade 4
* contraindication of ibuprofen (bleeding diasthesis, platelet count 10,000/mm3 or less, serum creatinine 2.0 mg/dL or greater, necrotizing enterocolitis stage 2 or greater

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe bronchopulmonary dysplasia (BPD) or mortality at 36 weeks postmenstrual age (PMA) | 36 weeks PMA

SECONDARY OUTCOMES:
Incidence of moderate to severe BPD | 36 weeks PMA
Incidence of oxygen dependency at 40 weeks PMA | 40 weeks PMA
Mortality rate | 28-days since birth and 36 weeks PMA
incidence of intraventricular hemorrhage (grade 3 or greater) | 28-days since birth
Incidence of retinopathy of prematurity (stage III or greater) | 40 weeks PMA (± 2 weeks)
Incidence of necrotizing enterocolitis (stage 2b or greater) | 40 weeks PMA (± 2 weeks)
Duration of PDA | 40 weeks PMA (± 2 weeks)
Duration of intubation | 36 weeks PMA
Duration of nasal continuous positive airway pressure (NCPAP) treatment | 40 weeks PMA (± 2 weeks)
Cumulative duration of oxygen use | 40 weeks PMA (± 2 weeks)
Incidence of adverse events | participants will be followed for the duration of hospital stay, an expected average of 12 weeks
Growth velocity | 40 weeks PMA (± 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Se In Sung, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung SI, Lee MH, Ahn SY, Chang YS, Park WS. Effect of Nonintervention vs Oral Ibuprofen in Patent Ductus Arteriosus in Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2020 Aug 1;174(8):755-763. doi: 10.1001/jamapediatrics.2020.1447. PMID 32539121